CLINICAL TRIAL: NCT06502366
Title: A Randomized, Placebo-controlled, Double-blind, Multicenter, 12-Week, 3-Way, Partial-replicate Crossover Pharmacodynamic Study to Assess the Equivalence of Budesonide and Albuterol (BDA) Delivered by MDI HFO Compared With BDA Delivered by MDI HFA in Participants With Asthma
Brief Title: A Study to Investigate the Effect on Lung Function of BDA Formulated With a Next Generation Propellant Compared With an Approved Asthma Treatment (BDA With HFA Propellant) in Participants With Asthma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6933C00002
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: This is a Randomized, Placebo-controlled, Double-blind, Multicenter, 12-Week, 3-Way, Partial-replicate Crossover Pharmacodynamic Study to Assess the Equivalence of BDA MDI HFO Compared with BDA MDI HFA in Participants with Asthma.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BDA MDI HFO (Active Comparator): 160/180 µg Budesonide/albuterol pressurized inhalation suspension, HFO
  Interventions: Drug: BDA MDI HFO 160/180 μg
- BDA MDI HFA (Active Comparator): 160/180 µg Budesonide/albuterol pressurized inhalation suspension, HFA
  Interventions: Drug: BDA MDI HFA 160/180 μg
- Placebo MDI HFA (Placebo Comparator): Placebo pressurized inhalation suspension, HFA
  Interventions: Drug: Placebo MDI HFA

INTERVENTIONS:
Drug: BDA MDI HFO 160/180 μg — Budesonide/albuterol pressurized inhalation suspension, HFO
  Arms: BDA MDI HFO
Drug: BDA MDI HFA 160/180 μg — Budesonide/albuterol pressurized inhalation suspension, HFA
  Arms: BDA MDI HFA
Drug: Placebo MDI HFA — Placebo pressurized inhalation suspension, HFA
  Arms: Placebo MDI HFA

SUMMARY:
The purpose of this study is to assess the PD equivalence of the approved asthma combination therapy, BDA, delivered using the proposed replacement propellant HFO compared with BDA delivered using the currently approved propellant HFA in participants with asthma.

DETAILED DESCRIPTION:
The purpose of this study is to assess the PD equivalence of the approved asthma combination therapy, BDA, delivered using the proposed replacement propellant HFO compared with BDA delivered using the currently approved propellant HFA in participants with asthma.

The study duration for each participant will be approximately 14 to 15 weeks and will consist of:

1. A screening and placebo run-in period of approximately 2 weeks prior to the first dose of study intervention
2. 3 treatment periods of 4 weeks each
3. A final safety follow-up visit via telephone contact approximately 5 days after the final dose of study intervention

Participants will attend in-clinic visits 2 weeks apart during the screening/run-in period (Visits 1 and 2) and then every 4 weeks during the treatment period (Visits 3, 4, and 5).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 years of age at the time of signing the ICF.
* Participants who have physician diagnosed asthma as defined by GINA for at least 12 months prior to Visit 1.
* Eligible participants are on either a) no daily inhaled maintenance therapy or b) daily inhaled maintenance therapy with low-dose ICS or low-dose ICS-LABA. Participants who are on low-dose ICS maintenance therapy are required to be stable on therapy for a minimum of 3 months prior to Visit 1; participants using low-dose ICSLABA maintenance regimens are required to be stable on therapy for a minimum of 6 months prior to Visit 1.
* Participants with a pre-bronchodilator FEV1 of ≥ 60% and < 90% predicted normal at Visit 1 or Visit 1a.
* Participants with a pre-dose FEV1 of ≥ 60% and < 90% predicted normal at Visit 2 that is within ± 20% of their Visit 1 pre-bronchodilator FEV1.
* Participants who demonstrate bronchodilator responsiveness defined as a > 12% and > 200 mL increase in FEV1 relative to baseline following administration of study provided SABA at Visit 1 or Visit 1a.
* Participants able to demonstrate acceptable spirometry performance as defined by the acceptability and repeatability criteria in the ATS/ERS Standardization of Spirometry 2019 update
* Participants who are willing and, in the opinion of the investigator, able to adjust current asthma therapy, as required by the protocol.
* Participants with a body mass index < 40 kg/m2.
* Females must not be of childbearing potential or, if of childbearing potential, using a form of birth control

Exclusion Criteria:

* Confirmed or suspected diagnosis of COPD or clinically significant non-asthma airway/lung disease.
* Systemic corticosteroid use (eg, prednisone for 3 or more days or a single depo-injectable dose of corticosteroids) for any respiratory, immune, or allergy-attributed disease within 6 months prior to Visit 1.
* An upper respiratory infection requiring antibiotic treatment that is not resolved within 7 days prior to Visit 1.
* A lower respiratory infection in the 4 weeks prior to Visit 1.
* Life-threatening asthma defined as any history of significant asthma episode(s) requiring admission to an intensive care unit, positive pressure ventilation associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma-related syncopal episode(s) within 5 years of Visit 1.
* Hospitalization due to asthma within 12 months or systemic corticosteroid usage (eg, prednisone for 3 or more days or a single depo-injectable dose of corticosteroids) for asthma within 6 months prior to Visit 1.
* A severe asthma exacerbation during the run-in period
* An ePRO device alert during the run-in period with investigator-confirmed worsening asthma symptoms
* Historical or current evidence of a clinically significant disease including, but not limited to: cardiovascular (eg, congestive heart failure, known aortic aneurysm, clinically significant cardiac arrhythmia, coronary heart disease), hepatic, renal, hematological, neuropsychological, endocrine (eg, uncontrolled diabetes mellitus, uncontrolled thyroid disorder, Addison's disease, Cushing's syndrome), or gastrointestinal (eg, poorly controlled peptic ulcer, gastroesophageal reflux disease) disorders. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the participant at risk through study participation or that could affect the efficacy or safety analyses if the disease/condition exacerbated during the study.
* Unresectable cancer that has not been in complete remission for at least 5 years prior to Visit 1
* Hospitalization for psychiatric disorder or attempted suicide within 1 year of Visit 1.
* Known history of drug or alcohol abuse within 12 months of Visit 1 or known abuse at any time during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2026-03-03 (Estimated); Study Completion 2026-03-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in peak FEV1 in 0-60 minutes after dosing at Day 29 | Change from baseline at Day 29
  To assess the equivalence of BDA MDI HFO relative to BDA MDI HFA on lung function in participants with asthma.
Change from baseline in peak FEV1 in 0-60 minutes after dosing at Day 29 | Change from baseline at Day 29
  To demonstrate assay sensitivity via superiority of BDA MDI HFA relative to placebo MDI HFA on lung function in participants with asthma

SECONDARY OUTCOMES:
Change from baseline in morning pre-dose trough FEV1 | Change from baseline at Day 29
  To assess the equivalence of BDA MDI HFO relative to BDA MDI HFA on lung function in participants with asthma.
Change from baseline in morning pre-dose trough FEV1 | Change from baseline at Day 29
  To demonstrate assay sensitivity via superiority of BDA MDI HFA relative to placebo MDI HFA on lung function in participants with asthma

CONTACTS AND LOCATIONS:
Locations (135):
- United States (73):
  - Research Site, Mobile, Alabama
  - Research Site, Sheffield, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Encinitas, California
  - Research Site, Fullerton, California
  - Research Site, Gardena, California
  - Research Site, Huntington Beach, California
  - Research Site, La Mesa, California
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, San Bernardino, California
  - Research Site, San Diego, California
  - Research Site, San Jose, California
  - Research Site, Santa Ana, California
  - Research Site, Stockton, California
  - Research Site, Van Nuys, California
  - Research Site, Westminster, California
  - Research Site, Englewood, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Boynton Beach, Florida
  - Research Site, Miami, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Rincon, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Meridian, Idaho
  - Research Site, River Forest, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Sioux City, Iowa
  - Research Site, Louisville, Kentucky
  - Research Site, Lafayette, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, White Marsh, Maryland
  - Research Site, Flint, Michigan
  - Research Site, Columbia, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Monticello, New York
  - Research Site, New York, New York
  - Research Site, Watertown, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Pottstown, Pennsylvania
  - Research Site, Scottdale, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, North Charleston, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Boerne, Texas
  - Research Site, Dallas, Texas
  - Research Site, DeSoto, Texas
  - Research Site, El Paso, Texas
  - Research Site, Kingwood, Texas
  - Research Site, McKinney, Texas
  - Research Site, Pearland, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Victoria, Texas
  - Research Site, West Jordan, Utah
  - Research Site, Burke, Virginia
  - Research Site, Portsmouth, Virginia
  - Research Site, Spokane, Washington
  - Research Site, Morgantown, West Virginia
  - Research Site, Milwaukee, Wisconsin
- China (31):
  - Research Site, Baotou
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chizhou
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Huizhou
  - Research Site, Jinan
  - Research Site, Jinhua
  - Research Site, Lanzhou
  - Research Site, Linhai
  - Research Site, Nanchang
  - Research Site, Pingxiang
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Taiyuan
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xuzhou
  - Research Site, Yangzhou
  - Research Site, Yinchuan
  - Research Site, Zhengzhou
  - Research Site, Zhuji
- Malaysia (6):
  - Research Site, Alor Star
  - Research Site, Ampang
  - Research Site, Cheras
  - Research Site, Petaling Jaya
  - Research Site, Rawang
  - Research Site, Sandakan
- Mexico (13):
  - Research Site, Chihuahua City
  - Research Site, Cuernavaca
  - Research Site, Culiacán
  - Research Site, Durango
  - Research Site, Guadalajara
  - Research Site, Mazatlán
  - Research Site, Mexico City
  - Research Site, Mérida
  - Research Site, Monterrey
  - Research Site, San Juan del Río
  - Research Site, Tijuana
  - Research Site, Veracruz
  - Research Site, Zapopan
- Thailand (4):
  - Research Site, Bangkoknoi
  - Research Site, Khon Kaen
  - Research Site, Mueang
  - Research Site, Ratchathewi
- Research Site, Abu Dhabi, United Arab Emirates
- United Kingdom (3):
  - Research Site, Ashton-under-Lyne
  - Research Site, Glasgow
  - Research Site, Newcastle upon Tyne
- Vietnam (4):
  - Research Site, Can Tho
  - Research Site, Haiphong
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/